CLINICAL TRIAL: NCT04981652
Title: Whole Milk to Augment Muscle Protein Synthesis in Older Women: a Randomized Controlled Trial
Brief Title: The Effect of Whole Milk to Improve Muscle Health in Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HIREB 4832
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Dairy Products; Muscle Protein Synthesis; Aging; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to one of three intervention groups (whole milk, skim milk or almond beverage)
Who Masked: Participant
Masking Description: Participant was blinded by formulating intervention beverages to have a similar taste profile with noncaloric, non-nutritional flavouring additives
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole Milk (Experimental): Participants randomly assigned to the whole milk condition will undergo three sequential study phases, each lasting three days in length. During phase 1, these participants will participate in habitual physical activity and consume a standardized diet, delivering 0.8 g/kg/body mass per day of protein. During the second phase, participants in this group will continue to perform habitual activity, but will have two whole milk experimental beverages (250 mL each serving, 3% milk fat) added to their standardized diet each day for the three day period. Finally, during the last three days of the study, participants will continue to consume the their intervention diet, but their physical activity levels (monitored via daily step count) will be increased to ~150% of their habitual levels.
  Interventions: Dietary Supplement: Whole Milk
- Skim Milk (Experimental): Participants randomly assigned to the skim milk condition will undergo three sequential study phases, each lasting three days in length. During phase 1, these participants will participate in habitual physical activity and consume a standardized diet, delivering 0.8 g/kg/body mass per day of protein. During the second phase, participants in this group will continue to perform habitual activity, but will have two skim milk experimental beverages (250 mL each serving, 0% milk fat) added to their standardized diet each day for the three day period. Finally, during the last three days of the study, participants will continue to consume the their intervention diet, but their physical activity levels (monitored via daily step count) will be increased to ~150% of their habitual levels.
  Interventions: Dietary Supplement: Skim Milk
- Almond Beverage (Experimental): Participants randomly assigned to the almond beverage condition will undergo three sequential study phases, each lasting three days in length. During phase 1, these participants will participate in habitual physical activity and consume a standardized diet, delivering 0.8 g/kg/body mass per day of protein. During the second phase, participants in this group will continue to perform habitual activity, but will have two almond experimental beverages (250 mL each serving) added to their standardized diet each day for the three day period. Finally, during the last three days of the study, participants will continue to consume the their intervention diet, but their physical activity levels (monitored via daily step count) will be increased to ~150% of their habitual levels.
  Interventions: Dietary Supplement: Almond Beverage

INTERVENTIONS:
Dietary Supplement: Whole Milk — Participants will consume twice daily whole milk beverages in addition to a standardized diet.
  Arms: Whole Milk
Dietary Supplement: Skim Milk — Participants will consume twice daily skim milk beverages in addition to a standardized diet.
  Arms: Skim Milk
Dietary Supplement: Almond Beverage — Participants will consume twice daily almond beverages in addition to a standardized diet.
  Arms: Almond Beverage

SUMMARY:
Muscle and strength begin to noticeably decline around 50 years of age, increasing an individual's risk for disease and disability. Although changes in muscle mass ultimately depend on the balance of muscle protein synthesis (MPS) and breakdown (MPB) of muscle proteins, the latter remains relatively constant with aging. Accordingly, interventions that increase rates of MPS may combat long-term decrements in skeletal muscle mass and function. Previous research has established that an optimal diet to maintain muscle mass in elderly individuals requires relatively large amounts of high-quality protein to be consumed at each meal of the day. While this is a seemingly simple strategy, there are some barriers to increasing protein feeding in elderly individuals, particularly the cost of high-quality protein and, sometimes, difficulty with chewing/swallowing. Moreover, older adults often do not wish to consume large portions of protein in one meal.

Milk is a readily accessible, affordable and nutritious source of nutrient-dense high-quality protein. Consuming milk with each meal is an easy strategy to promote the maintenance of skeletal muscle mass with aging. There is also evidence suggesting that a higher fat content of milk can have a beneficial role in stimulating the MPS response to feeding, but there are insufficient data to recommend this strategy to elderly individuals.

The primary aim is to measure the rates of MPS in response to controlled diets providing whole milk, fat-free milk, or a control supplement (almond beverage - often marketed as an 'alternative' to milk) with each meal. All diets will provide equal amounts of energy, but the dairy interventions will provide more protein, reflecting the amount of protein provided by each beverage. The investigators hypothesize that rates of MPS will be highest in the whole milk group but that fat-free milk will still elicit a greater MPS than almond beverage. The investigators will conduct the comparison of beverages under habitual physical activity levels and under a brief period of increased physical activity (i.e., increased daily steps). Thus, the investigators will be able to determine whether MPS responses to the experimental beverages are increased in combination with physical activity. The results will provide evidence regarding the effectiveness of daily milk ingestion for the maintenance of muscle in the elderly, increasing the marketability of milk, and potentially whole milk.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 60-75 years (inclusive)
* Be at least 5 years post-menopausal
* Have a body mass index (BMI) between 20-35 kg/m2
* Be able to maintain a habitual diet, physical activity patterns, and body mass throughout the trial
* Be in general good health
* Understand the study procedures and sign this form providing informed consent to participate in the study.
* Understand the study procedures and sign the form providing informed consent to participate in the study.

Exclusion Criteria:

* Use of tobacco or related products
* Use assistive walking devices (e.g., cane or walker)
* A history of neuromuscular problems or muscle and/or bone wasting diseases
* Any acute or chronic illness; cardiac, pulmonary, liver, or kidney abnormalities; insulin- or non-insulin-dependent diabetes or other metabolic disorders (all ascertained through medical questionnaires)
* Use of medications known to affect protein metabolism (i.e. corticosteroids, nonsteroidal anti-inflammatory drugs (prescription use or daily use of over the counter medication), or prescription strength acne medications)
* Use of anticoagulant medication
* History of statin myalgia
* Allergy to lactose or almonds
* Consuming a vegan diet

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Muscle Protein Synthesis | Assessed at baseline (day 0-3), intervention diet (4-7) and intervention diet + activity (day 8-10)
  Muscle protein synthesis will be calculated by determining the change in deuterated alanine enrichment in skeletal muscle proteins over each study phase

SECONDARY OUTCOMES:
Western Blotting | Assessed at baseline (day 0-3), intervention diet (4-7) and intervention diet + activity (day 8-10)
  The protein content of mechanistic target of rapamycin (mTOR) signalling components (i.e., mTOR, eIF4E-binding protein 1 (4EBP1), p70S6K and ribosomal protein S6 (rpS6) will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stokes T, Mei Y, Seo F, McKendry J, McGlory C, Phillips SM. Dairy and Dairy Alternative Supplementation Increase Integrated Myofibrillar Protein Synthesis Rates, and Are Further Increased when Combined with Walking in Healthy Older Women. J Nutr. 2022 Jan 11;152(1):68-77. doi: 10.1093/jn/nxab358. PMID 34610129